# Participation Trends in Bladder Cancer Clinical Trials - Exploring Engagement Dynamics Among Individuals Impacted by Bladder Cancer

An Informed Consent Form For Power Clinical Trial's Observational Study Patients With Bladder Cancer

Date: August 18, 2023

Navigating the Context of This Informed Consent Form

If you are in the process of completing this form, it signifies that you are being considered for participation in an observational clinical trial that specifically focuses on individuals grappling with bladder cancer. This form serves as a comprehensive manual, unveiling the study's overarching aims, intricate execution plan, and multifaceted implications, both positive and potentially otherwise. Engaging in thoughtful contemplation of your potential role prior to making a decision is of the utmost importance, and seeking counsel from a trusted advisor can provide invaluable insights. Should any intricacies of the information presented within this document remain unclear or if questions arise, rest assured that the researcher is readily available to provide necessary clarifications.

## Unveiling the Study's Objective

Bladder cancer is a type of cancer that originates in the cells lining the bladder, which is a hollow organ in the lower abdomen that stores urine produced by the kidneys. This cancer typically begins in the innermost layer of the bladder and can potentially spread to deeper layers or to other parts of the body.

Treatment for bladder cancer depends on various factors such as the stage and type of cancer, as well as the patient's overall health. Options may include surgery to remove

the tumor or the entire bladder (cystectomy), chemotherapy, radiation therapy, immunotherapy, and targeted therapy. Early detection and prompt medical intervention are important for improving outcomes and reducing the spread of disease.

Clinical trials addressing bladder cancer play a crucial role in evaluating the safety and effectiveness of innovative treatments for this condition. These trials are instrumental in determining whether these emerging treatments outperform existing options and provide substantial evidence to support their wider adoption.

This particular study places meticulous focus on delving into the experiences of individuals diagnosed with bladder cancer as they actively engage in a distinct clinical trial involving medical interventions. The primary emphasis lies in closely examining trial completion rates and instances of voluntary withdrawal among these participants.

#### Significance of Observational Studies

By joining this medical trial, you step into the realm of an observational study, a distinctive subset of clinical exploration meticulously designed to glean insights by observing individuals while keeping their care regimens intact.

Researchers will meticulously chart your progress and diligently evaluate the outcomes of your condition without any form of intervention. This intricate trial methodology serves as a cornerstone in elevating our understanding of the trajectory of a specific medical condition and its effects on the lives of those bearing its diagnosis. Your active participation in this observational study plays a pivotal role in advancing the frontiers of medical understanding and fostering refinements in the care provided to individuals who share the same medical journey.

# This Trial Compared to Other Bladder Cancer Clinical Trials

A crucial aspect to acknowledge is that the foundation of this clinical trial rests upon an observational paradigm, underscoring that your engagement will not involve the administration of specific treatments or interventions as part of the study. Nonetheless, bladder cancer clinical trials encompass a spectrum of variations. For example, interventional trials that may require participants to undergo specific treatment regimens. This study, on the other hand, is purely observational.

Crafting an informed decision regarding your potential participation in a clinical trial demands an active approach of exploration and comparison among various studies. A wealth of information concerning <u>studies revolving around bladder cancer</u> can be readily accessed through platforms such as clinicaltrials.gov. Additionally, Power's dedicated online platform serves as a comprehensive repository of ongoing <u>bladder cancer clinical trials</u> that actively seek participants. By engaging in diligent research and cultivating a holistic understanding of diverse clinical trial formats, you empower yourself to confidently shape your path of participation.

## **Engaging Willingly in Clinical Trial Surveys**

Within the scope of this observational clinical trial, we cordially invite you to share your experiences with us. This endeavor entails your periodic completion of questionnaires every two weeks, a commitment estimated to consume approximately 20-30 minutes of your valuable time. Additionally, at quarterly intervals, we will arrange check-in calls, extending as long as your engagement with the trial persists.

It is pivotal to emphasize that your involvement in the survey phase of the trial hinges solely upon your discretion. The prerogative to decide whether to respond to specific queries or all inquiries lies entirely with you, and you retain the autonomy to conclude your participation in the trial at any juncture of your choosing. We wholeheartedly recognize that the decision to partake in a clinical trial is inherently personal, and our unwavering commitment is dedicated to furnishing the support you may require. Your privacy and comfort stand as paramount considerations, and we are unwavering in our commitment to honor your decision-making journey throughout the course of the trial.

# Ensuring the Privacy of Your Answers

Preserving the complete confidentiality of your information ranks among our highest priorities throughout the course of this clinical trial. With the aim of safeguarding your anonymity, we respectfully request that you refrain from incorporating any personal or identifiable particulars when responding to the questionnaires. The unwavering dedication of our research team is geared towards reinforcing the protective shield surrounding your confidentiality. Nevertheless, it is vital to acknowledge that specific legal scenarios may surface, compelling the release of your data.

#### Potential Risks

While clinical trials undeniably drive medical progress, it is crucial to recognize the potential presence of health risks that may loom over participants, especially in trials exploring novel treatments.

Nevertheless, our observational clinical trial departs from the norm by proactively alleviating this concern. We avoid subjecting participants to new interventions, effectively minimizing the risk. Instead, our core emphasis centers on observation and measuring outcomes, ensuring the absence of undue health hazards.

### Potential Advantages

Although immediate advantages might not be immediately evident for individuals partaking in this observational clinical trial, their participation carries the potential to create a meaningful impact on the lives of others. The repository of data amassed from participants will drive the enhancement of future protocols for enrolling patients with bladder cancer, potentially expanding access to medical research pathways. By undertaking this clinical voyage, individuals have the opportunity to catalyze transformative change within the realm of medical research, potentially altering the course for future bladder cancer patients.

Embarking on an In-Depth Exploration of Clinical Trial Inclusivity

For those who nurture a curiosity to read about representation within clinical trials, a wealth of online resources eagerly awaits your active engagement.

Whether your objective is to understand or simply to enrich your personal journey through the realm of clinical trials, these sources of knowledge stand as a guide:

Camidge, D. Ross, Haeseong Park, Karen E. Smoyer, Ira Jacobs, Lauren J. Lee, Zemfira Askerova, Justin McGinnis, and Yousef Zakharia. "Race and ethnicity representation in clinical trials: findings from a literature review of Phase I oncology trials." *Future Oncology* 17, no. 24 (2021): 3271-3280.

<u>Yates, Isabelle, Jennifer Byrne, S. Donahue, Linda McCarty, and Allison Mathews.</u>
<u>"Representation in clinical trials: A review on reaching underrepresented populations in research." *Clinical Researcher* 34, no. 7 (2020).</u>

#### Confirmation of Informed Assent

I hereby confirm that I have dedicated significant time to comprehensively understand and internalize the contents encapsulated within the informed consent form, either through self-directed exploration or with the guidance of a trusted individual who has conveyed its essence to me. All inquiries and reservations that occupied my thoughts have been diligently addressed to my complete satisfaction.

I am well aware that my participation in this study is a result of my voluntary decision, and the right to retract my consent resides solely with me, devoid of any obligation to furnish justification or assume financial commitments. I have been explicitly informed that a duplicate of this informed consent form will be furnished for my personal records.

Having conscientiously pondered and evaluated the entirety of the information presented to me, I hereby express my agreement to partake in this study, signifying my autonomous and informed choice.

| Printed Name of Participant |
|-----------------------------|
| • |
| Participant Signature |
| Tartiolparit Olgridiano |
| Date |

Validation by Informed Consent Facilitator

I affirm with confidence that I have engaged in a thorough dialogue with the participant, systematically elucidating the intricacies enfolded within this textual composition. My objective was to ensure the participant's comprehensive understanding of the trial's overarching aims, methodologies employed, potential risks and benefits, along with other pivotal aspects inherent to the bladder cancer clinical trial.

Ample opportunity was granted to the participant, encouraging the emergence of inquiries and facilitating the clarification of uncertainties or misconceptions. It is of utmost importance to underscore that the participant's involvement in this trial is a direct outcome of their voluntary decision, and they retain the unrestricted prerogative to discontinue their participation at any juncture, driven by any rationale, without encountering any financial burdens.

Following the participant's provision of consent, a meticulously preserved duplicate of this textual document was furnished to them, serving as a repository for their individual records.

| Printed Name of Person Taking Consent |
|---------------------------------------|
| Signature of Person Taking Consent |
| Date |